CLINICAL TRIAL: NCT05467280
Title: Women's Involvement in Steady Exercise (WISE) Project
Brief Title: WISE Project - Women's Involvement in Steady Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Collaborators: European Commission (Other); European Platform for Sport Innovation (Unknown); University Union - Nikola Tesla (Unknown); European Culture and Sport Organization (Unknown); Kinetic Analysis (Unknown); SPORTLAB S.S.D.A.R.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1944476
Record Dates: First submitted 2022-06-29; First posted 2022-07-20 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-06

CONDITIONS: Sedentary Lifestyle; Physical Inactivity
Keywords: Sedentary Behaviors
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): They will be given HIIT exercise video sessions twice a week for 6 months, through a mobile application where they will also be given nutritional and health advice, webinars, and challenges.
  Interventions: Other: Online HIIT Intervention
- Control (No Intervention): They will not carry out any type of intervention, they will only be monitored during the 6 months

INTERVENTIONS:
Other: Online HIIT Intervention — They will be given HIIT exercise video sessions twice a week for 6 months, through a mobile application where they will also be given nutritional and health advice, webinars and challenges.
  Arms: Intervention

SUMMARY:
The general objective is to assess adherence to a HIIT-type exercise program, complemented with nutritional plans and other health-related advice, which will be administered through a mobile application in sedentary girls.

DETAILED DESCRIPTION:
The project is aimed at encouraging participation in sport and physical activity, especially by supporting the implementation of the Council Recommendation on health-enhancing physical activity and being in line with the EU Physical Activity Guidelines, since its main objective is to determine the influence of exercise and healthy lifestyle on body composition of young women aged 15-24 and to define a specific WISE Exercise Programme - a multidimensional model of dependence between body composition, lifestyle and nutrition which would enable the programming of optimal patterns of behaviour in life habits as a planned corrective measure and stimulate the young women in EU countries to avoid the drop out of sports.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 15 and 24 years.
2. Sedentary participants who do not comply with the WHO physical exercise recommendations and with a low IPAQ, which means that they do not perform at least:

   * 3 or more days of vigorous activity for at least 20 minutes a day.
   * 5 or more days of moderate-intensity activity.
   * Walk at least 30 minutes a day every day.
   * 5 or more days of combined moderate or vigorous intensity activities or walking achieved a minimum of 600 METs(min/week).

Exclusion Criteria:

1. Participants with diabetes.
2. Participants with possible heart problems or other type of contraindication that does not allow physical exercise (for this, the PAR-Q survey will be passed)
3. Participants who are not willing to wear the watch during the 6 months that the intervention lasts.
4. Participants who have contracted severe COVID-19 in the last 3 months. If the patients suffer from COVID-19 during the study, then they will stop exercising, but the measurements will be taken at the end of the study.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 281 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in daily steps from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Measured as the daily step count assessed via the Xiaomi Mi Band 5

SECONDARY OUTCOMES:
Adherence (Asistence) | T2 (6 months)
  Exercise diary, asking the participants if they have completed the exercise each session
Adherence (Retention) | T2 (6 months)
  Number of participants who are still following the WISE exercise videos or the follow-up measurements
Adherence (Duration) | T2 (6 months)
  Number of participants who had done a minimum of 20 minutes of exercise two times a week.
Adherence (Intensity) | T2 (6 months)
  Exercise diary, asking the participants their perceived exertion of the sessions via the modified Borg Scale after they just done it. The Borg Rating of Perceived Exertion is a way of measuring physical activity intensity level. A 0-10 scales is used where 0 is no perceived exertion (rest) and 10 is maximal perceived exertion.
Change in body weight (kg) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Assessment of body weight (kg) is conducted using bioelectrical impedance analysis with the multi frequency segmented body composition analyzer InBody 230 (InBodyUSA, Cerritos, CA).
Change in skeletal muscle mass (kg) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Assessment of skeletal muscle mass (kg) is conducted using bioelectrical impedance analysis with the multi frequency segmented body composition analyzer InBody 230 (InBodyUSA, Cerritos, CA).
Change in body fat mass (kg) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Assessment of body fat mass (kg) is conducted using bioelectrical impedance analysis with the multi frequency segmented body composition analyzer InBody 230 (InBodyUSA, Cerritos, CA).
Change in body mass index (BMI) (kg/m2) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Assessment of BMI (kg/m2) is conducted using bioelectrical impedance analysis with the multi frequency segmented body composition analyzer InBody 230 (InBodyUSA, Cerritos, CA).
Change in core strength (plank test) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Messured in seconds via the plank test protocol
Change in endurance (6 minutes walking test) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Meters
Change in the international Physical Activity Questionnaire (IPAQ) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  The IPAQ assesses walking and activities of a moderate and vigorous intensity that are per-formed continuously for at least 10 min in all domains of everyday life (i.e. leisure, occupa-tional, household and transport) in the last 7 days.
Change in the Health Lifestyle and Personal Control Questionnaire (HLPCQ) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  This is a 26-item tool in which the respondent is asked to indicate the frequency of adopting 26 positively stated lifestyle habits using a Likert-type scale (1 = Never or rarely, 2 = Sometimes, 3 = Often and 4 = Always)
Change in the physical Activity Enjoyment Scale from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Is an 18-item scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7- point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it)
Change in period pain (hours) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Total hours of pain the participants has during their period
Change in period pain (intensity) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Pain intensity will be measured using the visual analogue scale (VAS). A 100-millimeter line bounded by ''no pain'' on the left (0) and ''worst pain possible'' (100) on the right will be used to indicate the average pain during the period.
Change in the Pittsburgh Sleep Quality Index (PSQI) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Change in conditioned pain modulation (CPM) from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Assessment of CPM in clinical practice can document the (in)efficacy of the endogenous anti-nociceptive system. we analyzed the effect that CPM had through the cold pressure test and pressure pain thresolds of the quadriceps
Change in cold pain threshold from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  The second when the participant sense pain in the cold pressor test.
Change in cold pain inensity from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Level of pain brought on by the cold water on a 0 to 10 numerical rating scale (NRS), where 0 is regarded as no pain and 10 is the most agonizing pain imaginable. Measured just before the hand is removed from the water in the cold pressor test
Cold pain tolerance from baseline to 3 and 6 months | T0(Baseline), T1 (3 months) and T2 (6 months)
  Second where the girls take the hand out of the water container in the cold pressor test

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de Valencia, Valencia, Spain